CLINICAL TRIAL: NCT02652858
Title: Central and Peripheral Arterial Pressure Decoupling In Cardio-Pulmonary Bypass
Acronym: CAPD-CPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Université Joseph Fournier Grenoble 1 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL15_0400
Record Dates: First submitted 2016-01-06; First posted 2016-01-12 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cardiopulmonary Bypass; Cardiac Surgery; Extracorporeal Circulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulse wave's speed observational arm (Experimental): Whole patients for who the pulse wave's speed are measured during a cardiopulmonary bypass during cardiac surgery
  Interventions: Procedure: Non-invasive blood pressure oscillometer (NIBP) implementation

INTERVENTIONS:
Procedure: Non-invasive blood pressure oscillometer (NIBP) implementation — Implementation of two additional NIBP on humeral and femoral sites.

SUMMARY:
Central and peripheral arterial pressure decoupling occurs in some clinical conditions like sepsis or cardiopulmonary bypass. This decoupling may leed to unsuitable decisions such as the use of catecholamines.

The aim of this study is to evaluate the pulse wave's speed as a marker of central and peripheral arterial pressure decoupling in a scheduled condition which is the cardiopulmonary bypass during cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled patient for coronary or valvular surgery with cardiopulmonary bypass
* Cardiopulmonary bypass is at least 90 minutes
* Written consent is needed

Exclusion Criteria:

* Patient with heart rate disorder
* Patient with aortic dissection
* Dobutamine/milrinone/levosimendan treatment before surgery
* Patient with heart rate due to a pacemaker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Measurement of femoral, radial and humeral pulses during a cardiopulmonary by-pass (CPBP). | Day one (6 times)
  Pulse wave's speed is calculated using 1) time between ECG R-wave and local detection of the pulse wave (femoral, humeral and radial) 2) a length from heart to these sites.
  Wave detection at femoral and humeral sites will use oscillometry and wave detection at radial site will use an invasive catheter which is always set for this surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] N. Smal, L. Guigue, D. Anglade, C. Lavault, F. Grimbert, Y. Lavault, F. Boucher, J.L. Fellahi. Assessment of central-peripheral arterial pressure decoupling: a preliminary study in cardiac surgery under cardiopulmonary bypass (CPB). Abstract presented at the Annual Congress of the French Society of Anaesthesia and Intensive Care (SFAR), Paris, 2017.